CLINICAL TRIAL: NCT00288054
Title: A Pilot (Phase I) Study of Weekly Docetaxel and Cetuximab Chemoradiation for Poor Risk Stage III Non-Small Cell Lung Cancer
Brief Title: S0429: Docetaxel, Cetuximab, and Radiation Therapy in Treating Patients With Stage III Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study closed early due to poor accrual.
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000456381; U10CA032102 (NIH); S0429 (Other: SWOG)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2012-12-25 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; large cell lung cancer; squamous cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung | interventions — Cetuximab; Docetaxel; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cetuximab + Radiotherapy (no Docetaxel) (Experimental)
  Interventions: Biological: cetuximab; Radiation: radiation therapy
- Cetuximab + Radiotherapy + Docetaxel (Experimental)
  Interventions: Biological: cetuximab; Drug: docetaxel; Radiation: radiation therapy

INTERVENTIONS:
Biological: cetuximab — Cohorts 1 and 2: 400 mg/m2 (initial dose) 2 hour IV infusion on Day 1, Cycle 1 only.
  250 mg/m2, 1 hour IV infusion on Days 8 , 15 and 22 during Cycle 1. 250 mg/m2 (subsequent doses), 1 hour IV infusion on Days 1, 8 , 15 and 22 during subsequent cycles.
Drug: docetaxel — Cohort 2 ONLY: 20 mg/m2 IV over 15 - 30 minutes on Days 8, 15 and 22 of Cycle 1. Concurrent with RT and cetuximab starting at Week 2.
  20 mg/m2 IV over 15 - 30 minutes on Days 1, 8, 15 and 22 of Cycle 2.
  Arms: Cetuximab + Radiotherapy + Docetaxel
Radiation: radiation therapy — Radiation therapy should begin on Day 8 of Cycle 1 and continue through the end of Cycle 2. Refer to Section 12.1 for Radiation Therapy Review.
  RT prescription should be PTV (GTV + 2-cm margins on CT scan) to 6,480 cGy in 36 fractions given 5 days a week, 180 cGy per day. The dose is prescribed to the isocenter. The entire treatment should be planned prior to starting treatment to ensure that the plan meets protocol specifications.

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some find tumor cells and kill them or carry tumor-killing substances to them. Others interfere with the ability of tumor cells to grow and spread. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving docetaxel and cetuximab together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel when given together with cetuximab and radiation therapy in treating patients with stage III non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Test the feasibility and toxicity of combined cetuximab, weekly docetaxel, and concurrent radiotherapy in patients with poor-risk stage III non-small cell lung cancer (NSCLC).

Secondary

* Evaluate response rates (confirmed and unconfirmed, complete and partial) as well as overall and progression-free survival.
* Correlate EGFR mutations, KRAS mutations, EGFR/HER2 gene copy number detected by FISH, and protein expression by immunohistochemistry of EGFR-HER signaling pathways, phosphorylation, proliferative markers, apoptotic markers, selected oncogene markers, and markers for angiogenesis in biopsied pre-treatment tumor tissues with response and survival outcomes.
* Explore possible associations between changes in plasma angiogenic factors (VEGF, IL-8, bFGF) and cytokine levels (IL-6, IL-1α, ICAM, TGF-β, and others) and the risk of treatment-related pneumonitis and esophagitis.

OUTLINE: Patients are enrolled sequentially to 1 of 2 treatment groups.

* Cohort 1: Patients receive cetuximab IV over 1-2 hours on days 1, 8, 15, and 22.
* Cohort 2: Patients receive cetuximab as in group 1 followed by docetaxel IV over 15-30 minutes on days 8, 15, and 22 of course 1 and on days 1, 8, 15, and 22 of course 2.

Initially, 27 patients will be enrolled in Cohort 1. Once all patients in Cohort 1 have discontinued treatment, if toxicity rates are acceptable per protocol specifications, an additional 27 patients will be enrolled to Cohort 2. Treatment in both cohorts repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity. All patients also undergo radiotherapy once daily, 5 days a week, beginning on day 8 of course 1 and continuing through course 2 (approximately 7 weeks). Patients with no progressive disease then receive cetuximab alone once weekly. Treatment with cetuximab alone continues in the absence of disease progression for up to 2 years.

After completion of study treatment, patients are followed periodically for up to 3 years.

PROJECTED ACCRUAL: A total of 54 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically proven newly diagnosed single, primary, bronchogenic stage IIIA or selected stage IIIB (excluding malignant pleural effusion) non-small cell lung cancer (NSCLC) of one of the following cellular types:

  * Adenocarcinoma
  * Large cell carcinoma
  * Squamous cell carcinoma
  * Unspecified
* Histology or cytology from involved mediastinal or supraclavicular nodes will be sufficient for diagnosis if a separate primary lesion of the lung parenchyma is clearly evident on radiographs (i.e., a second biopsy will not be required)
* Underwent positron emission tomography (PET) scan within the past 42 days

  * N2 or N3 mediastinal disease by PET scan OR enlarged nodes on CT scan determined to be N2 or N3 by biopsy
* Measurable disease, defined as lesions that can be accurately measured in at least one dimension as ≥ 2 cm by conventional techniques or ≥ 1 cm by spiral CT scan

  * Pleural effusion, ascites, bone lesions, and laboratory parameters are not considered measurable disease
* No brain metastases
* Malignant pleural effusion allowed provided 1 of the following is true:

  * Present before mediastinoscopy or exploratory thoracotomy AND the pleural fluid is transudate with negative cytology
  * Present only after but not before exploratory or staging thoracotomy AND the pleural fluid is either transudate or exudate with negative cytology
  * Present only on CT scan but not on decubitus chest x-ray AND deemed too small to tap under either CT scan or ultrasound guidance

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1, meeting ≥ 1 of the following criteria OR Zubrod performance status 2 with no co-morbidities or meeting 1 of the following criteria:

  * No co-morbidities
  * FEV_1 < 2 L OR < 1 L with estimated contralateral FEV_1 ≥ 0.6 L
  * DLCO > 10 mL/mm Hg/min
  * Albumin < 0.85 times lower limit of normal
  * Unintentional weight loss > 10% within the past 6 months
  * Controlled congestive heart failure which, in the opinion of the investigator, may become decompensated due to radiotherapy
* FEV_1 < 2 L OR < 1 L with estimated contralateral FEV_1 ≥ 0.6 L
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Must provide prior smoking history
* Serum bilirubin normal
* Meets one of the following criteria:

  * Alkaline phosphatase (AP) ≤ 4 times ULN AND SGOT or SGPT normal
  * AP normal AND SGOT or SGPT ≤ 2.5 times ULN
* No other prior malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or adequately treated stage I or II cancer from which the patient is currently in complete remission
* No pregnant or nursing patients
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or curative surgery for this cancer
* No prior radiotherapy to the neck and/or thorax for any reason
* No prior therapy which specifically targets the EGFR pathway
* No concurrent growth factors (e.g., filgrastim [G-CSF], epoetin alfa, or pegfilgrastim) or amifostine
* No concurrent intensity-modulated radiotherapy
* No concurrent prophylactic mediastinal, contralateral hilar, or supraclavicular lymph node radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuhchyau Chen, MD, PhD, Principal Investigator — James P. Wilmot Cancer Center; Kishan J. Pandya, MD, Principal Investigator — James P. Wilmot Cancer Center; Derick H. Lau, MD, Principal Investigator — University of California, Davis; Karen Kelly, MD, Principal Investigator — University of Colorado, Denver; Laurie E. Gaspar, MD, MBA, Principal Investigator — University of Colorado, Denver
Locations (77):
- United States (77):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Tibotec Therapeutics - Division of Ortho Biotech Products, LP, Marysville, California
  - University of California Davis Cancer Center, Sacramento, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Regional Cancer Center, Edwards, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Valley View Hospital Cancer Center, Glenwood Springs, Colorado
  - Montrose Memorial Hospital Cancer Center, Montrose, Colorado
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - West, Boca Raton, Florida
  - Eugene M. and Christine E. Lynn Cancer Institute at Boca Raton Community Hospital - Main Campus, Boca Raton, Florida
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Hematology Oncology Consultants - Naperville, Naperville, Illinois
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Caritas St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Good Samaritan Cancer Center at Good Samaritan Hospital, Kearney, Nebraska
  - Tucker Center for Cancer Care at Orange Regional Medical Center, Middletown, New York
  - Highland Hospital of Rochester, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Danville Regional Medical Center, Danville, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: Cetuximab + Radiotherapy (no Docetaxel): Eligible patients who began protocol treatment were included in the analysis.
Period: Overall Study
Arm/Group | Cohort 1: Cetuximab + Radiotherapy (no Docetaxel)
Started | 24
Completed | 0
Not Completed | 24
Not completed — Protocol Violation | 2
Not completed — Lack of Efficacy | 16
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Not protocol specified | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cohort 1: Cetuximab + Radiotherapy (no Docetaxel)
Number analyzed (Participants) | 22
Age Continuous [Median (Full Range); unit: years] | 72 [51 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Secondary Outcome: Toxicity
Description: Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Weekly for the first 8 weeks, then every 4 weeks while subject on protocol treatment.
Population: Eligible patients who received protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Cetuximab + Chest Radiation Therapy
Number analyzed (Participants) | 22
Participants
  Allergic reaction/hypersensitivity | 1
  Ataxia (incoordination) | 1
  Burn | 1
  Cardiac troponin I (cTnI) | 1
  Cough | 1
  Dehydration | 1
  Diarrhea | 1
  Dyspnea (shortness of breath) | 3
  Esophagitis | 1
  Fatigue (asthenia, lethargy, malaise) | 1
  Hypoxia | 1
  Inf (clin/microbio) w/Gr 3-4 neuts - Lung | 1
  Left ventricular diastolic dysfunction | 1
  Lymphopenia | 4
  Magnesium, serum-low (hypomagnesemia) | 3
  Muscle weakness, not d/t neuropathy - Extrem-lower | 1
  Neurology-Other (Specify) | 1
  Neutrophils/granulocytes (ANC/AGC) | 1
  Pain - Head/headache | 1
  Pain - Skin | 1
  Potassium, serum-low (hypokalemia) | 1
  Rash: acne/acneiform | 2
  Syncope (fainting) | 1
  Thrombosis/thrombus/embolism | 1

2. Primary Outcome: Treatment-related Esophagitis or Pneumonitis
Description: The primary endpoint will be the rate of Grade 3 or greater esophagitis and/or pneumonitis within 4 months after discontinuation of radiation therapy.
Time Frame: Weekly for the first 8 weeks, then every 4 weeks thereafter for up to 4 months after complettion of radiotherapy.
Population: Eligible patients who received protocol treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Cetuximab + Radiotherapy (no Docetaxel)
Number analyzed (Participants) | 22
percentage of participants | 5 [0 to 23]

3. Secondary Outcome: Overall Survival
Description: The duration form the date of enrollment until the date of death due to any cause. Patients last known to be alive are censored at the date of last contact.
Time Frame: weekly while patient is on protocol treatment, then monthly thereafter.
Population: Eligible patients who began protocol treatment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Cetuximab + Radiotherapy (no Docetaxel)
Number analyzed (Participants) | 22
months | 14 [8 to 24]

4. Secondary Outcome: Progression-free Survival.
Description: Duration from the date of enrollment until the date of progression (as defined by RECIST: >= 20% increase over baseline in the sum of longest diameters, or appearance of new lesions, or non-measurable disease that is clearly worsening in the opinion of the treating investigator, or symptomatic deterioration) or death due to any cause. Patients last known to be alive and free of disease progression are censored at the date of last contact.
Time Frame: At week 10, week 22, and then every 3 months until progression for up to 3 years after enrollment.
Population: Eligible patients who began protocol treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: Cetuximab + Radiotherapy (no Docetaxel)
Number analyzed (Participants) | 22
months | 8 [5 to 9]

5. Secondary Outcome: Response Rate
Description: Confirmed and unconfirmed complete and partial responses in the subset of patients with measurable disease (as defined per RECIST). A confirmed complete response (CR) is defined as disappearance of all disease, confirmed by a second determination of CR at least 4 weeks later. A confirmed partial response (PR) is defined as a >= 30% decrease from baseline in the sum of longest diameters, confirmed by a second determination of PR at least 4 weeks later. A patient is considered to have measurable disease if they have at least one lesion with a longest diameter of >= 2 cm by conventional CT, or >= 1 cm by spiral CT.
Time Frame: Week 10 and week 22
Population: Eligible patients who began protocol treatment and who had measurable disease (as defined by RECIST) at baseline were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Cetuximab + Radiotherapy (no Docetaxel)
Number analyzed (Participants) | 19
percentage of participants | 47 [24 to 71]

ADVERSE EVENTS:
Time Frame: Weekly for the first 8 weeks, then every 4 weeks while on protocol treatment.
Arm/Group | Cetuximab + Chest Radiation Therapy
Serious Adverse Events (participants affected / at risk) | 5/22
Other Adverse Events (participants affected / at risk) | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Chest Radiation Therapy (N=22)
Left ventricular diastolic dysfunction (Cardiac disorders) | 1
Inf (clin/microbio) w/Gr 3-4 neuts - Lung (Infections and infestations) | 2
Cardiac troponin I (cTnI) (Investigations) | 1
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 1
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1
Adult respiratory distress syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab + Chest Radiation Therapy (N=22)
Hemoglobin (Blood and lymphatic system disorders) | 8
Cardiac-ischemia/infarction (Cardiac disorders) | 2
SVT and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 3
SVT and nodal arrhythmia - Sinus tachycardia (Cardiac disorders) | 4
Ocular/Visual-Other (Specify) (Eye disorders) | 3
Vision-blurred vision (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 9
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 10
Esophagitis (Gastrointestinal disorders) | 9
Heartburn/dyspepsia (Gastrointestinal disorders) | 5
Hemorrhoids (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 3
Pain - Esophagus (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Constitutional Symptoms-Other (Specify) (General disorders) | 2
Edema: limb (General disorders) | 5
Fatigue (asthenia, lethargy, malaise) (General disorders) | 15
Fever in absence of neutropenia, ANC lt1.0x10e9/L (General disorders) | 3
Pain-Other (Specify) (General disorders) | 2
Allergic reaction/hypersensitivity (Immune system disorders) | 4
Inf w/normal ANC or Gr 1-2 neutrophils - Skin (Infections and infestations) | 2
Inf w/normal ANC or Gr 1-2 neutrophils - UTI (Infections and infestations) | 2
Infection-Other (Specify) (Infections and infestations) | 2
Opportunistic inf associated w/gt=Gr 2 lymphopenia (Infections and infestations) | 2
Bruising (in absence of Gr 3-4 thrombocytopenia) (Injury, poisoning and procedural complications) | 3
Burn (Injury, poisoning and procedural complications) | 2
Rash: dermatitis associated w/Chemoradiation (Injury, poisoning and procedural complications) | 3
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 3
AST, SGOT (Investigations) | 3
Alkaline phosphatase (Investigations) | 4
Creatinine (Investigations) | 2
INR (of prothrombin time) (Investigations) | 2
Leukocytes (total WBC) (Investigations) | 2
Lymphopenia (Investigations) | 7
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 2
Platelets (Investigations) | 2
Weight gain (Investigations) | 2
Weight loss (Investigations) | 4
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 6
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 3
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 8
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 2
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 6
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 2
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 3
Muscle weakness, not d/t neuropathy - Extrem-lower (Musculoskeletal and connective tissue disorders) | 4
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 2
Pain - Back (Musculoskeletal and connective tissue disorders) | 4
Pain - Chest wall (Musculoskeletal and connective tissue disorders) | 3
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 2
Pain - Joint (Musculoskeletal and connective tissue disorders) | 2
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2
Pain - Neck (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 3
Neurology-Other (Specify) (Nervous system disorders) | 2
Neuropathy: sensory (Nervous system disorders) | 2
Ocular/Visual-Other (Specify) (Nervous system disorders) | 3
Pain - Head/headache (Nervous system disorders) | 2
Taste alteration (dysgeusia) (Nervous system disorders) | 3
Mood alteration - depression (Psychiatric disorders) | 2
Pain - Bladder (Renal and urinary disorders) | 2
Urinary frequency/urgency (Renal and urinary disorders) | 3
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 10
Hemorrhage, pulmonary/upper respiratory - Lung (Respiratory, thoracic and mediastinal disorders) | 2
Hemorrhage, pulmonary/upper respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 6
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 2
Dermatology/Skin-Other (Specify) (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4
Nail changes (Skin and subcutaneous tissue disorders) | 2
Pain - Skin (Skin and subcutaneous tissue disorders) | 2
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 15
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No